CLINICAL TRIAL: NCT06342609
Title: Effect of Colchicine on Progression of Known Coronary Atherosclerosis in Patients With STable CoROnary Artery Disease CoMpared to Placebo - EKSTROM Trial
Brief Title: Effect of Colchicine on Progression of Known Coronary Atherosclerosis in Patients With Stable Coronary Artery Disease
Acronym: EKSTROM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Responsible Party: Principal Investigator, Matthew J. Budoff, Investigator, Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: 32857-01-EKSTROM
Record Dates: First submitted 2024-03-16; First posted 2024-04-02 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Double blind Placebo controlled
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Colchicine (Active Comparator): 0.5 milligram (mg) per day of Colchicine orally administered over the period of 52 weeks
  Interventions: Drug: Colchicine 0.5 MG
- Placebo (Placebo Comparator): 0.5mg per day of Placebo orally administered over the period of 52 weeks
  Interventions: Drug: Colchicine 0.5 MG

INTERVENTIONS:
Drug: Colchicine 0.5 MG — 0.5mg per day of Colchicine orally administered
  Other Names: Mitigare; Colcrys

SUMMARY:
This is a randomized double-blind, placebo-controlled, investigator-initiated trial that compares Colchicine 0.5mg/day with placebo, among patients with stable CAD. Subjects will be educated to maintain medication compliance with other prescribed medications.

DETAILED DESCRIPTION:
The goal of this study is to evaluate whether treatment with Colchicine results in greater change of low attenuation plaque volume from baseline level when compared to placebo in subjects with stable Coronary Artery Disease (CAD). The Primary objective of the study is to determine progression rates of low attenuation plaque under influence of Colchicine as compared to placebo. The study will also look to determine effects of Colchicine on the morphology and composition non -calcified coronary plaque, progression of total plaque volume, progression of high vulnerability features of plaque and to assess whether these effects are modulated by a change in HsCRP and other markers of inflammation (HsCRP, IL-6, IL-1α, IL-1β, IL-18) as well as the effect on Pericoronary adipose tissue (PCAT) and Epicardial adipose tissue (EAT) volume and well as on the endothelial function.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30-85 years
2. Proven coronary artery disease; as evidenced by coronary angiography, CT coronary angiography or a Coronary Artery Calcium Score (Agatston score >400).
3. Clinically stable for at least six months
4. Patients should have no major competing co-morbidities or contra-indication to colchicine therapy
5. Patients must be considered to be compliant with their usual therapy
6. Willingness to be on birth control for women of childbearing age or established postmenopausal for at least 1 year
7. Patients must provide written informed consent after the scope and nature of the investigation has been explained to them.
8. Patients must be considered to be compliant with their usual therapy
9. Patients must provide written informed consent after the scope and nature of the investigation has been explained to them.
10. Patients must be able and willing to comply with the requirements of this study protocol

Exclusion Criteria:

1. Women who are pregnant, breast feeding or may be considering pregnancy during the study period
2. Renal impairment as evidenced by a serum creatinine >150 μmol/l or estimated glomerular filtration rate (eGFR) <50mL/min/1.73m2
3. Severe heart failure - systolic or diastolic New York Heart Association Functional classification 3 or 4
4. Moderate or severe valvular heart disease considered likely to require intervention
5. Dependency, frailty or a predicted life expectancy < 5 years
6. Peripheral neuritis, myositis or marked myo-sensitivity to statins
7. Requirement for long term colchicine therapy for any other reason
8. Current enrollment in another trial
9. Patients with inflammatory bowel disease (Crohn's disease or ulcerative colitis) or patients with chronic diarrhea
10. Any unstable medical, psychiatric or substance abuse disorder that in the opinion of the investigator or principal investigator is likely to affect the subject's ability to complete the study or precludes the subject's participation in the study
11. Patient with progressive neuromuscular disease of Creatine Phosphokinase (CPK) level >3 times the upper limit of normal as measured within the past 30 days and determined to be non-transient through repeat testing.
12. Patients already taking long term colchicine therapy for any other reason
13. History of malignancy within the last 5 years (other than skin cancer) or evidence of active cancer which would require concomitant cancer chemotherapy
14. Hematological or biochemical values at screening outside the reference ranges considered as clinically significant in the opinion of the investigator or PI.
15. Allergy to contrast material

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2023-03-15 (Actual); Primary Completion 2024-09-07 (Actual); Study Completion 2024-09-07 (Actual)

PRIMARY OUTCOMES:
Rate of change in low attenuation plaque volume as measured by multidetector computed tomography (MDCT) angiography | 12 months
  Reduction of low attenuation plaque volume from baseline (start of the study) till the final visit will be measured using Coronary Computed Tomography Angiography (CTA).

SECONDARY OUTCOMES:
Effect of Colchicine on markers of inflammation using laboratory tests | 12 months
  To determine the effect of Colchicine on markers of inflammation (IL-6, IL-1α, IL-1β, IL-18 high sensitivity C-reactive protein)
Effects of Colchicine on Pericoronary Adipose Tissue (PCAT) volume using CTA | 12 months
  To determine the effects of Colchicine on PCAT volume.
Effects of Colchicine on Epicardial Adipose Tissue (EAT) volume using CTA | 12 months
  To determine the effects of Colchicine on EAT volume.
Effect of Colchicine on the markers of Endothelial Function using Flow-mediated dilation (FMD) | 12 months
  To determine the effect of Colchicine on Endothelial function using FMD.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Budoff, MD, Principal Investigator — The Lundquist Institute
Locations (1):
- Lundquist Institute for Biomedical Innovation at Harbor UCLA Medical Center, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Budoff MJ, Bhandari M, Iskander B, Ghanem AK, Kinninger A, Stark J, Garikapati V, Chilukuri S, Hankil V, Krishnan S, Punnanithinont N, Ichikawa K, Kambalapalli S, Hamal S, Lakshmanan S. Effect of colchicine on progression of known coronary atherosclerosis in patients with stable coronary artery disease: EKSTROM randomized placebo controlled trial. Eur Heart J Cardiovasc Imaging. 2026 Feb 11:jeag028. doi: 10.1093/ehjci/jeag028. Online ahead of print. PMID 41670023
- [Derived] Verghese D, Hamal S, Ghanem A, Kinninger A, Javier D, Ichikawa K, Benzing T, Krishnan S, Kianoush S, Hamidi H, Bagheri M, Abraham D, Deljavanghodrati M, Ghoto A, Aldana-Bitar J, Budoff M. Effect of colchicine on progression of known coronary atherosclerosis in patients with STable CoROnary artery disease CoMpared to placebo (EKSTROM) trial-rationale and design. Am Heart J. 2024 Nov;277:20-26. doi: 10.1016/j.ahj.2024.07.005. Epub 2024 Jul 17. PMID 39029568